CLINICAL TRIAL: NCT07388862
Title: Comparison of Treatment Outcome of Pulpotomy With Versus Without Dental Operating Microscope in Carious Mature Permanent Teeth : A Randomized Controlled Trial
Brief Title: Comparison of Treatment Outcome of Pulpotomy With Versus Without Dental Operating Microscope in Carious Mature Permanent Teeth
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Sirawut Hiran-us, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBC 28/2025
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy; treatment outcome; dental operating microscope

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional using of dental operating microscope in the procedure (Experimental): using of dental operating microscope in the procedure for improving the quality of treatment
  Interventions: Device: Dental operating microscope
- Routine pulpotomy (No Intervention): Routine pulpotomy procedure without addition using of dental operating microscope

INTERVENTIONS:
Device: Dental operating microscope — Incorperating the using of dental operating microscope into the pulpotomy procedure
  Arms: Additional using of dental operating microscope in the procedure

SUMMARY:
The goal of this [randomized clinical trial] is to evaluate the treatment outcome by assessing clinical and radiographic outcomes.

The main question it aims to answer is

Do using dental operating microscope incorperated with pulpotomy procedure will have a different outcome when compare with without using.

Participants will be asked to have clinical and radiographic evaluation for evaluating the outcome every year after treatment.

DETAILED DESCRIPTION:
Materials and methods Study design and setting This study is a prospective, single-center, single-blinded, parallel-group, randomized controlled trial conducted at the Dental Department, Phaholponpayuhasena Hospital. All clinical procedures are performed by a single experienced endodontist. Clinical outcome evaluations are carried out by the same operator, while radiographic outcome evaluations are conducted by another experienced endodontist.

Study participants Inclusion Criteria

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent teeth diagnose with asymptomatic or symptomatic irreversible pulpitis. Diagnoses are confirmed using EPT and cold tests. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013)20.
* Teeth are restorable with direct composite restoration. Exclusion Criteria
* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening
* Bleed cannot be stopped within 8 minutes after full pulpotomy21,22

Treatment procedure A comprehensive medical and dental history is taken before treatment. Preoperative data, including age, sex, tooth number are recorded in a predesigned patient's chart. The treatment, the study design, alternative treatment modalities, potential benefits, risks, and follow-up protocol are explained to the qualifying patients and informed consent is obtained from the voluntary patients who are willing to participate in the study.

Sample size calculation The sample size calculation is based on a suspected difference of 39.2% in the success rate between the control and magnification group in MB2 orifice finding using n4Studies with a 5% α error. The minimum sample size was calculated to be 46. Considering patients lost to follow-up, a total of 50 teeth from different patients are included in this study.

Randomization and masking Block randomization with variable 4 block sizes is used to generate a sequence of random numbers for allocating the patients equally into two study groups. Each random blocks are sealed in an opaque envelope which is opened at the beginning of the clinical trial by the operator. New block will be open after all the patient in the previous block was completed and repeat until the end of the clinical trials to ensure the equality of group distribution: The vital pulp therapy with and without magnification intervention groups.

Intervention All the treatment is carried out by a single operator. All the patients received a topical anesthesia before local anesthesia. An inferior alveolar nerve block (1.8 ml 2% Lidocaine with epinephrine 1:100,000)+buccal infiltration (1.7 ml 4% Articaine with epinephrine 1:100,000) for mandibular teeth, buccal infiltration (1.8 ml 2% Lidocaine with epinephrine 1:100,000) for maxillary teeth. The anesthesia is confirmed by negative response to EPT. The pulpotomy procedure is performed under rubber dam isolation in a single visit. If the patient experienced pain during the procedure, an additional anesthesia is used to achieve profound pulpal anesthesia by intraligament injection with 0.3 ml 2% Lidocaine with epinephrine 1:100,000. The operating field is disinfected with iodine and alcohol. A cylindrical diamond airotor operates under air water coolant to outline the cavity. Low speed round bur and a spoon excavator are used to remove the soft carious dentine using nonselective caries removal from the periphery towards the centre of the carious lesion. The deepest layer of carious dentine is thereafter disinfected with 2 ml of 2.5% NaOCl prior to pulpal exposure.

The patient will have his or her eyes covered with a dental drape and randomly divided into the following two groups:

Group I (Magnification) : The remaining procedures will be carried on under Zeiss OPMI Pico dental operating microscope (Carl Zeiss Meditec, Germany) with total magnification ranging from 3.6× to 6.0×. More aspects will be included in this group which included:

* If the remaining resected pulp is avascular with necrotic or yellowish liquefied areas, or microscopic hemostasis cannot be achieved, then further tissue removal is attempted
* Ensure the absence of dentin chips and blood clotting above remaining pulp tissue.
* Complete removal of detached pulp tissue and dentine fragments into a vascular pulp.

Group II (Control) : The remaining procedures will be carried on under naked eye.

The new high-speed sterile diamond airotor is used to completely remove the coronal pulp tissue. Then direct passive irrigation with of 2.5% NaOCl solution up to 8 minutes to arrest the bleeding. The time to achieve hemostasis is recorded in minutes and seconds. The diagnosis of vital inflamed pulp is confirmed by the presence of bleeding in the pulp chamber.

In both study groups, 1 mm calcium silicate cement putty type (Totalfil-ERRM) is placed as a caping agent over the residual pulp.The tooth is restored with Resin Modified Glass Ionomer Cement (RMGIC) base (Vitrebond, 3M) and composite restoration (Z350XT, 3M) and polishing in the same visit.

The full pulpotomy cases where bleeding from residual pulp cannot be arrested within 8 minutes, are excluded from the study, and pulpectomyare performed. Immediate post-operative periapical radiograph is taken.

Treatment outcome assessment All the teeth are assessed clinically at 6 months and every year and radiographs are taken. Clinically asymptomatic teeth without any radiographic evidence of periapical rarefaction or root resorption are categorized as success in strict criteria and categorized as survival in loose criteria when clinically asymptomatic teeth with periapical rarefaction.

Recall Clinical evaluation and periapical radiograph will be taken. The quality of the coronal restoration is checked, and the restorations are repaired if deemed necessary. In case of failed cased, the cause of failure will be identified and recorded. Proper treatment will be proposed for specific problem.

Clinical evaluation included

* Coronal restoration
* EPT
* Percussion
* Palpation
* Mobility
* Probing depth
* Occlusion All clinical evaluation will be evaluated by the same operator who was blinded from the intervention.

Radiographic evaluation included

* Periapical radiograph The same operator will judge the quality of the recall radiograph which include
* 3x3 mm area covered the periapical area
* No distortion or blurred
* The image is able to interpret the periapical tissue

The blinded experienced endodontist will be evaluate the radiographic success of recall radiograph by recording as:

* Normal periapical tissue
* Thickening PDL space
* Periapical lesion

Statistical analysis The Kolmogorov-Smirnov test is used to assess the normality of continuous data. Fisher's exact test analyze demographic variables. The dichotomous outcome of success versus failure will be used as the dependent variable to statistically analyze the prognostic factors. The impact of prognostic factors on treatment outcomes will be statistically analyzed using bivariate and multivariate multilevel logistic regression. Success rates between groups are analyzed using the t-test. A p-value of < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent teeth diagnose with asymptomatic or symptomatic irreversible pulpitis. Diagnoses are confirmed using EPT and cold tests. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013)20.
* Teeth are restorable with direct composite restoration.

Exclusion Criteria:

* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening
* Bleed cannot be stopped within 8 minutes after full pulpotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-21 (Estimated); Primary Completion 2036-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome | Yearly up to 10 years
  Treatment outcomes will be classified as healed, healing, or failure based on clinical and radiographic evaluations.
  Healed: Cases presenting with no clinical symptoms and no evidence of a periapical lesion on radiographic examination.
  Healing: Cases presenting with no clinical symptoms and a reduction in the size of the periapical lesion on radiographic examination.
  Failure: Cases presenting with clinical symptoms and/or enlargement of the periapical lesion on radiographic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Sirawut Hiran-us, Study Director — Faculty of Dentistry, Chulalongkorn University; Choontawee Soponsakulkaew, Principal Investigator — Phaholponpayuhasena Hospital

IPD SHARING:
Plan to Share IPD: Undecided